CLINICAL TRIAL: NCT00846950
Title: Effects of H1-Antagonist on Stages of Human Information Processing
Brief Title: Effects of H1-Antagonist on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Effects of H1-antagonist on stages of human information processing, Dr. A. Vermeeren
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 06-3-075
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Cognition
Keywords: H1-antagonist; Event Related Potentials; Memory; Information processing; The effects of an H1 antagonist (dexchlorpheniramine) on human cognition
MeSH Terms: interventions — dexchlorpheniramine; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Drug: dexchlorpheniramine, lorazepam

INTERVENTIONS:
Drug: dexchlorpheniramine, lorazepam

SUMMARY:
The purpose of this study is to determine whether histamine is involved in memory and specific processes in human cognition.

DETAILED DESCRIPTION:
The neurotransmitter histamine appears to be involved in human cognitive performance. However, the exact role is very unclear. The role it plays in memory performance is highly disputed, as animal studies show decreased performance when the H1-receptor is blocked in the central nervous system while such findings in humans is scarce. To clarify the role of histamine in human memory and different processes in cognition, the effects of an H1-antagonist (dexchlorpheniramine) on memory, alertness and sensory and motor processes are measured. The study will be conducted according to a within subject cross-over design using healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a physician

Exclusion Criteria:

* present or history of any neurological of psychiatric disease
* present or history of any substance abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
P300 latency and LRP onset latency | 1.5 hours after treatment

SECONDARY OUTCOMES:
Words recalled | 1.5 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Vermeeren, Ph.D., Principal Investigator — Maastricht University hospital
Locations (1):
- Faculty of Psychology and Neuroscience, Maastricht University, Maastricht, Limburg, Netherlands